CLINICAL TRIAL: NCT02319096
Title: Whole Body Vibration Plate Therapy and Pelvic Floor Muscle Strength in Females With Stress Urinary Incontinence
Brief Title: Vibration Training and Pelvic Floor Muscle Strength in Females With Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medway NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Professor Jonathan Duckett, Consultant Obstetrician and Gynaecologist, Medway NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedwayNHS
Record Dates: First submitted 2014-10-15; First posted 2014-12-18 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Urinary Stress Incontinence
Keywords: Whole body vibration therapy; pelvic floor muscle training; stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with stress incontinence (Experimental): Patients who present to urogynaecology clinic with proven stress urinary incontinence who will be offered Whole body vibration therapy.
  Interventions: Other: Whole body vibration therapy

INTERVENTIONS:
Other: Whole body vibration therapy — Whole body vibration therapy using the Galileo machine as therapy for pelvic floor muscle training

SUMMARY:
Pelvic floor muscle training (PFMT) is the first line therapy recommended by NICE for the treatment of SUI. Due to poor motivation and compliance only 15-20% of women comply with the regimen. Whole body vibration (WBV) exercise has been developed as a new modality in the field of physiotherapy. The Galileo machine is a unique device for applying whole-body vibration. The investigators are currently using this therapy as an alternative to traditional pelvic floor muscle therapy. The investigators aim to audit the investigators treatment of whole body vibration.

DETAILED DESCRIPTION:
Pelvic floor muscle training (PFMT) is the first line therapy recommended by NICE for the treatment of SUI. It was first described by Arnold Kegel almost 60 years ago. PFMT exercises help the patient strengthen the muscles of the pelvic floor by the repeated high-intensity, rapid pelvic muscle contractions of both slow and fast twitch muscle fibres. The training of these muscles is difficult particularly when women have trouble in the perception of their PFM. This results in poor motivation and compliance with a Cochrane review suggesting that only 15-20% of women comply with the regimen.

Whole body vibration (WBV) exercise has been developed as a new modality in the field of physiotherapy. Whole body vibration (WBW) has a positive effect on muscle strength and rate of force. Stochastic WBV causes up to 12 muscle contractions per second which cannot be achieved by routine PFM exercise with supervision of a physiotherapist. The Galileo machine is a unique device for applying whole-body vibration. The investigators aim to audit their treatment of whole body vibration. This would be done using the patient global impression of improvement scale (PGI-I) and routine quality of life and symptoms questionnaires (International Consultation on Incontinence Female lower Urinary Tract Symptoms Questionnaire -ICIQ-FLUTS and Pelvic Floor Distress Inventory - PFDI) to be completed by the patient at initial appointment and 12 weeks after treatment and pelvic floor muscle assessment carried out at initial appointment and at 12 weeks. Patients will also have a qualitative interview with the Urogynaecology team to assess if therapy was found to be suitable and acceptable to patients.

ELIGIBILITY:
Inclusion Criteria:

1. Stress predominant urinary incontinence
2. Female patients >18 years

Exclusion Criteria:

1. Urgency predominant urinary incontinence
2. Symptomatic pelvic organ prolapse requiring intervention
3. Patients with bladder pathology (eg haematuria of unknown origin, UTI)
4. Contraindication to Whole Body Vibration

   * Musculoskeletal

     * Hip or knee endoprosthesis
     * Acute disc herniation
     * Joint fusion with metal implants
     * Acute arthritis
     * Osteoporosis with vertebral fracture
     * Recent Fracture
     * Acute Soft Tissue Injury
     * Acute Rheumatoid Arthritis
   * Cardiovascular

     * Recent myocardial infarction
     * Hypertension
     * Serious cardiovascular disease
     * Artificial heart valves
     * Pacemaker
     * Venous Thrombosis
     * Aortic Aneurysm
     * Peripheral vascular disease
     * Untreated orthostatic hypotension
     * Hernia
   * Neuromuscular

     * Impaired sensation
     * Impaired cognition
     * Deep brain and spinal cord stimulators
   * Other

     * Malignant tumours
     * Acute oedema
     * Impaired skin integrity of foot or leg
     * Recent surgery
     * Severe diabetes or migraines
     * Kidney and bladder stones
     * Pregnancy
     * Recently placed intrauterine devices or pins

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Patient Global Impression of Improvement scale (PGI-I) | 12 weeks
  Patients will be asked answer the PGI-I questionnaire after a full 12 week course of therapy

SECONDARY OUTCOMES:
International Consultation on Incontinence Female lower Urinary Tract Symptoms Questionnaire | 12 weeks
  Patients will be asked to answer the ICIQ-FLUTS to assess symptom improvement after a full 12 week course of therapy
Pelvic Floor Distress Inventory - PFDI | 12 weeks
  Patients will be asked to answer the PFDI-I to assess any improvement in quality of life after a full 12 weeks
Qualitative interview | 12 weeks
  A qualitative interview will be conducted with the urogynaecology team to assess if patients found the new therapy suitable and acceptable.
Pelvic muscle contraction | 12 weeks
  Pelvic muscle contraction will be measured at Week 0 and Week 12 using a pelvic perineometer to assess any improvement in pelvic muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan RA Duckett, FRCOG, Principal Investigator — Medway Maritime Hospital NHS Trust
Locations (1):
- Medway Maritime Hospital, Gillingham, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goode PS, Burgio KL, Locher JL, Roth DL, Umlauf MG, Richter HE, Varner RE, Lloyd LK. Effect of behavioral training with or without pelvic floor electrical stimulation on stress incontinence in women: a randomized controlled trial. JAMA. 2003 Jul 16;290(3):345-52. doi: 10.1001/jama.290.3.345. PMID 12865375
- [Result] Rovner ES, Wein AJ. Treatment options for stress urinary incontinence. Rev Urol. 2004;6 Suppl 3(Suppl 3):S29-47. PMID 16985862
- [Result] Luginbuehl H, Lehmann C, Gerber R, Kuhn A, Hilfiker R, Baeyens JP, Radlinger L. Continuous versus intermittent stochastic resonance whole body vibration and its effect on pelvic floor muscle activity. Neurourol Urodyn. 2012 Jun;31(5):683-7. doi: 10.1002/nau.21251. Epub 2012 Mar 6. PMID 22395850
- [Result] Kawanabe K, Kawashima A, Sashimoto I, Takeda T, Sato Y, Iwamoto J. Effect of whole-body vibration exercise and muscle strengthening, balance, and walking exercises on walking ability in the elderly. Keio J Med. 2007 Mar;56(1):28-33. doi: 10.2302/kjm.56.28. PMID 17392595
- [Result] Vella M, Nellist E, Cardozo L, Mastoroudes H, Giarenis I, Duckett J. Does self-motivation improve success rates of pelvic floor muscle training in women with urinary incontinence in a secondary care setting? Int Urogynecol J. 2013 Nov;24(11):1947-51. doi: 10.1007/s00192-013-2115-x. Epub 2013 May 24. PMID 23702666